CLINICAL TRIAL: NCT03337035
Title: The Effects of Probiotics and Oxytocin Nasal Spray on Social Behaviors of ASD Children- A Pilot Study
Brief Title: Probiotics and Oxytocin Nasal Spray on Social Behaviors of Autism Spectrum Disorder (ASD) Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Xuejun Kong,MD, Research Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017P001667
Record Dates: First submitted 2017-10-31; First posted 2017-11-08 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Probiotics, Oxytocin
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Phase 1: a. oral placebo, and b. oral probiotics; Phase 2: a. intranasal OXT + oral placebo, and b. intranasal OXT + oral probiotics
Who Masked: Participant, Care Provider, Investigator
Masking Description: this study will be double blinded for both participants/guardians and medication administrator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- oral probiotics and oxytocin spray (Active Comparator): Subjects will receive oral probiotics, 2 pills per day, for 28 weeks. For the last 12 weeks, subjects will also receive intranasal oxytocin spray at the following dose: 4 IU in week 1, 8 IU in week 2, 16 IU in week 3, and 24 IU in weeks 4-12.
  Interventions: Drug: intranasal oxytocin; Dietary Supplement: oral probiotics
- oral placebo and oxytocin spray (Placebo Comparator): Subjects will receive oral placebo, 2 pills per day, for 28 weeks. For the last 12 weeks, subjects will also receive intranasal oxytocin spray at the following dose: 4 IU in week 1, 8 IU in week 2, 16 IU in week 3, and 24 IU in weeks 4-12.
  Interventions: Drug: intranasal oxytocin; Dietary Supplement: oral placebo

INTERVENTIONS:
Drug: intranasal oxytocin — 4-24 IU per day, dosage gradually increases
  Other Names: Novartis Syntocinon
Dietary Supplement: oral probiotics — 200 million cfu per day
  Arms: oral probiotics and oxytocin spray
Dietary Supplement: oral placebo — 2 pills per day
  Arms: oral placebo and oxytocin spray

SUMMARY:
Because oral probiotics reported to potentially induce endogenous Oxytocin, and Oxytocin has been reported to improve social behaviors, the investigators will conduct a pilot trial to compare the effects of probiotics and Oxytocin on social behavioral changes in ASD children. Additionally, the investigators will check oxytocin levels, and perform brain fMRI in some subjects, in order to determine which treatment is more efficient, sustainable, and practical, and whether both treatments in combination are better than either treatment alone. If the trial is conclusive, the investigators will conduct a trial in large scale to understand more the mechanism of ASD behaviors and corresponding effective interventions.

DETAILED DESCRIPTION:
This study description is in accordance with the Consolidated Standards of Reporting Trials (CONSORT) guidelines that are published for the evaluation of randomized controlled trials. This clinical trial is a randomized, double-blind placebo controlled study. Subjects will be randomized to 2 groups:

Phase 1: a. oral placebo, and b. oral probiotics; Phase 2: a. intranasal Oxytocin(OXT) + oral placebo, and b. intranasal OXT + oral probiotics

The treatment will proceed for a total of 28 weeks. In the first phase (16 weeks), all the patients will be randomly and proportionally divided into two groups: Group A (30 subjects) receives oral probiotics while Group B (30 subjects) receives an oral placebo. In the second phase, subjects in Group A and Group B will continue their respective oral probiotics or placebo administration as in Phase 1. In addition, both groups will be simultaneously administered with intranasal OXT spray.

Testing will be performed 3 times total (before, during, and after treatment). The tests include behavioral surveys, cognitive tests, clinical autonomic tests, and blood tests for oxytocin levels. Investigators plan to select up to 10 subjects from each group to conduct a series of MRI studies at week 0, week 16 and week 28.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 3-25years old;
2. Pre-existing diagnosis of autism; subjects may be asked to provide documentation confirming diagnosis by DSM-V-TR criteria, ADOS, ADI-R, or other clinical forms
3. A care provider who can reliably bring the participant to study visits;
4. No planned changes in medications or psychosocial interventions during trial (stable medications within the last 2 weeks);
5. Willingness to provide blood samples

Exclusion Criteria:

1. Pregnant woman (before or during the study).
2. Comorbidity of other neurological and/or psychiatric disorders such as unstable seizures, schizophrenia, schizoaffective disorder, bipolar disorders or history of substance abuse.
3. Psychotropic medication use
4. Subjects with active cardiovascular disease that is not controlled by medication.
5. Oxytocin, antibiotic, or probiotic use within the last 30 days.
6. Regular nasal obstruction or nosebleeds
7. Significant hearing, vision, or motor impairments
8. Habitual consumption of large volumes of water
9. Started taking new medications within the last 2 weeks

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Social Responsiveness Scale (SRS) Edition 2 | change from baseline at 0, 16, and 28 weeks
  social communication and behavior - The scoring is based on T-score which is based on the sum of responses as follows (76 to higher - severe, 66 to 75- moderate deficiencies, 60 to 65 - mild deficiencies, 59 and below is not clinically significant for ASD).
Aberrant Behavior Checklist (ABC) Edition 2 | change from baseline at 0, 16, and 28 weeks
  social behavior test - The total score is calculated based on 5 sub-scales (Irritability, Social Withdrawal, Stereotypic Behavior, Hyperactive/Noncompliance, and Inappropriate Speech). There are 58 questions that are scored on a 0-3 scale 0 -"not at all a problem", 1- "the behavior is a problem but slight in degree", 2- "the problem is moderately serious" and 3- "the problem is severe in degree". Based on this sub-scores are calculated and added to get the total score.

SECONDARY OUTCOMES:
Neuroinflammation and Oxytocin levels | change from baseline at 0, 16, and 28 weeks
  neuroendocrine biomarker measured in blood ( Melatonin, Oxytocin, Tumour Necrosis Factor alpha, testosterone and Interleukin 6)
structural MRI | change from baseline at 0, 16, and 28 weeks
  The software Freesurfer will be used to calculate volume of brain regions and diffusion parameters (e.g. fractional anisotropy and mean diffusivity) from structural T1 and diffusion tensor images respectively. T-tests will be applied for group comparisons.
Functional MRI (resting state) | change from baseline at 0, 16, and 28 weeks
  Correlation analysis will be used to calculate the connectivity across different brain regions. T-tests will be used for group comparisons.
Functional MRI (task based) | change from baseline at 0, 16, and 28 weeks
  General linear modeling will be used to calculate brain responses to the tasks. T-tests will be used for group comparisons.
Autonomic indices 1 | change from baseline at 0, 16, and 28 weeks
  Blood volume pulse
Autonomic indices 2 | change from baseline at 0, 16, and 28 weeks
  heart rate
Autonomic indices 3 | change from baseline at 0, 16, and 28 weeks
  peripheral skin temperature
Autonomic indices 4 | change from baseline at 0, 16, and 28 weeks
  skin electrodermal activity
Autonomic indices 5 | change from baseline at 0, 16, and 28 weeks
  blood oxygen saturation
Microbiome | change from baseline at 0, 16, and 28 weeks
  16s metagenomic sequencing of the microbiome
Eye tracking and Behavioral task (joint attention) | change from baseline at 0, 16, and 28 weeks
  joint attention - Conduct T-tests and calculate P values for total and average fixation values for each area of interest
Eye tracking and behavioral task (emotion response) | change from baseline at 0, 16, and 28 weeks
  emotion response - The accuracy and reaction time will be calculated for each time point. Then an ANOVA will be used to compare the results.
Eye tracking and behavioral task (eye behavior) | change from baseline at 0, 16, and 28 weeks
  eye behavior - Conduct T-tests and calculate P values for total and average fixation values for each area of interest

CONTACTS AND LOCATIONS:
Overall Officials: Xue-Jun Kong, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data with researchers not involved in this study.

REFERENCES:
- [Derived] Sherman HT, Liu K, Kwong K, Chan ST, Li AC, Kong XJ. Carbon monoxide (CO) correlates with symptom severity, autoimmunity, and responses to probiotics treatment in a cohort of children with autism spectrum disorder (ASD): a post-hoc analysis of a randomized controlled trial. BMC Psychiatry. 2022 Aug 8;22(1):536. doi: 10.1186/s12888-022-04151-3. PMID 35941573
- [Derived] Kong XJ, Liu J, Li J, Kwong K, Koh M, Sukijthamapan P, Guo JJ, Sun ZJ, Song Y. Probiotics and oxytocin nasal spray as neuro-social-behavioral interventions for patients with autism spectrum disorders: a pilot randomized controlled trial protocol. Pilot Feasibility Stud. 2020 Feb 12;6:20. doi: 10.1186/s40814-020-0557-8. eCollection 2020. PMID 32082606